CLINICAL TRIAL: NCT00842023
Title: A Randomized Controlled Trial to Evaluate Renal Function, Inflammatory Mediators, and Neurohormonal Markers in Acutely Decompensated Heart Failure Patients Receiving Nesiritide Compared to Nitroglycerin.
Brief Title: Assessment of Biomarkers and Cardiorenal Syndrome in Acute Decompensated Heart Failure With Vasodilator Therapy
Acronym: ABC-HFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Principal Investigator, Sheryl Chow, Associate Professor, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCP-26060
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Natriuretic peptides; BNP; Heart Failure; Nitoglycerin; Biomarkers
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nesiritide Infusion (Experimental): Nesiritide: 2 mcg/kg bolus (optional) followed by 0.01 mcg/kg/min infusion for 48 hours.
  Interventions: Drug: Nesiritide
- Nitroglycerin Infusion (Active Comparator): Nitroglycerin was initiated at 10 mcg/min initial starting dose titrated every 5-10 minutes until symptom relief, SBP<or= 90 mm Hg, or up to a maximum rate of 200 mcg/min plus standard treatment.
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nesiritide — Bolus 2 mcg/kg followed by 0.01 mcg/kg/min
  Arms: Nesiritide Infusion
Drug: Nitroglycerin — 5-10 mcg/min titrating per protocol based on blood pressure
  Arms: Nitroglycerin Infusion

SUMMARY:
The purpose of this study is to determine whether Nesiritide is more effective than nitroglycerin in modifying inflammatory and neurohormonal biomarkers without renal toxicity when proper infusion duration is administered.

DETAILED DESCRIPTION:
No additional details provided

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Subject must be able to understand the potential risks and benefits associated with the study.
* Baseline systolic blood pressure ≥ 90 mm Hg at the time of enrollment.
* Clinical symptoms of dyspnea and laboratory admission BNP levels > 500 pg/mL.
* Neither pregnant or breastfeeding at the time of enrollment.
* Authorization of patient's enrollment by patient's medical provider.

Exclusion Criteria:

* <18 years of age
* Denies written informed consent
* Pregnant or lactating.
* Baseline systolic BP < 90 mmHg or cardiogenic shock
* No symptoms of congestion or admission BNP < 500 pg/mL
* Known allergy to E.coli-derived products, or any history of anaphylactic reactions to nesiritide.
* Receiving dialysis at the time of enrollment.
* Serum creatinine > 2.5 mg/dL at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl L. Chow, PharmD, FCCP, BCPS, Principal Investigator — Western University of Heatlh Sciences
Locations (1):
- Centinela Hospital Medical Center, Inglewood, California, United States

REFERENCES:
- [Result] Chow SL, O'Barr SA, Peng J, Chew E, Pak F, Quist R, Patel P, Patterson JH, Heywood JT. Renal function and neurohormonal changes following intravenous infusions of nitroglycerin versus nesiritide in patients with acute decompensated heart failure. J Card Fail. 2011 Mar;17(3):181-7. doi: 10.1016/j.cardfail.2010.10.005. Epub 2010 Dec 3. PMID 21362524
- [Result] Chow SL, O'Barr SA, Peng J, Chew E, Pak F, Quist R, Patel P, Patterson JH, Heywood JT. Modulation of novel cardiorenal and inflammatory biomarkers by intravenous nitroglycerin and nesiritide in acute decompensated heart failure: an exploratory study. Circ Heart Fail. 2011 Jul;4(4):450-5. doi: 10.1161/CIRCHEARTFAILURE.110.958066. Epub 2011 May 16. PMID 21576282

RESULTS

PARTICIPANT FLOW:
Groups:
- Nesiritide Infusion: 2 mcg/kg bolus (optional) followed by 0.01 mcg/kg/min infusion for 48 hours.
- Nitroglycerin Infusion: 10 mcg/min initial starting dose titrated every 5-10 minutes until symptom relief, SBP<or= 90 mm Hg, or up to a maximum rate of 200 mcg/min plus standard treatment.
Period: Overall Study
Arm/Group | Nesiritide Infusion | Nitroglycerin Infusion
Started | 45 | 44
Completed | 45 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesiritide Infusion | Nitroglycerin Infusion | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 24 | 43
  >=65 years | 26 | 20 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 68.6 (14.1) | 66.8 (17.2) | 67.7 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants] — Sample size was estimated at 90 patients total; however, 1 patient was enrolled twice. Therefore, only 89 patients were enrolled in the primary study.
  participants
    United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Renal Function by Serum Creatinine
Description: Serum creatinine values and changes in serum creatinine
Time Frame: Baseline, 24 hours, 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Nesiritide: 2 mcg/kg bolus (optional) followed by 0.01 mcg/kg/min infusion for 48 hours.
- Nitroglycerin: 10 mcg/min initial starting dose titrated every 5-10 minutes until symptom relief, SBP<or= 90 mm Hg, or up to a maximum rate of 200 mcg/min plus standard treatment
Arm/Group | Nesiritide | Nitroglycerin
Number analyzed (Participants) | 45 | 44
mg/dL
  Serum creatinine at baseline | 1.3 (0.4) | 1.3 (0.4)
  Serum creatinine at 24 hours | 1.3 (0.4) | 1.4 (0.4)
  Serum creatinine at 48 hours | 1.3 (0.4) | 1.4 (0.5)

2. Other Pre Specified Outcome: Inflammatory Markers
Description: Interleukin-6
Time Frame: 48 hours
Population: Only participants with available data were assessed for this outcome measure.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Nesiritide Infusion | Nitroglycerin Infusion
Number analyzed (Participants) | 36 | 30
pg/mL | 25 (7) | 50 (5)

3. Other Pre Specified Outcome: Serum Levels of Cystatin-C
Description: Cystatin-C is a protease inhibitor and a sensitive endogenous marker of renal function.
Time Frame: Baseline, 24 hours, 48 hours
Population: Only participants with available data were assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nesiritide | Nitroglycerin
Number analyzed (Participants) | 36 | 30
ng/mL
  Cystatin-C at Baseline | 1332 (1308) | 2026 (1814)
  Cystatin-C at 24 Hours | 1475 (1291) | 3108 (3761)
  Cystatin-C at 48 Hours | 1449 (1298) | 2739 (3369)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Nesiritide Infusion | Nitroglycerin Infusion
Serious Adverse Events (participants affected / at risk) | 12/45 | 12/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nesiritide Infusion (N=45) | Nitroglycerin Infusion (N=44)
Symptomatic Hypotension (Cardiac disorders) | 5 (5) | 5 (5)
Death (General disorders) | 7 (7) | 7 (7) — Assessed at 6 months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes